CLINICAL TRIAL: NCT00843479
Title: The Aging Endocrine Pancreas: Characterization of the Entero-insular Axis Physiology in the Elderly.
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Bruno Geloneze, Dr. Bruno Geloneze, University of Campinas, Brazil
Other Study IDs: LIMED0006
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: diabetes mellitus, type 2; Insulin resistance; Aging; Incretins; DPP-IV protein, human; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide; insulin; glucagon; ghrelin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sera and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Elderly NGT: Normoglycemic subjects 65-80 years old
- Middle-age NGT: Middle-age normoglycemic subjects 35 to 50 years old.

SUMMARY:
Like most endocrine axes, the entero-insular axis is expected to go through an age-related physiological deterioration, what might contribute to special features of the elderly onset type 2 diabetes in comparison to middle-age.

Twenty four NGT volunteers will be evaluated by a meal tolerance test (MTT) for incretin hormone measurements, and by the hyperglycemic clamp followed by an arginine test for assessing the beta-cell function and the acute insulin response. Others parameters as body composition and basic biochemistry will be also evaluated at Laboratory of Investigation on Metabolism and Diabetes - LIMED / State university of Campinas, Brazil.

The characterization of the glucagon-like peptide-1 (GLP-1) production, dipeptidyl peptidase IV (DPP-IV) activity and/or endocrine pancreas incretin-response at aging, might be an interesting evidence to reinforce an incretin-based therapeutic approach for elderly onset type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Stable weight (< 5% variation) within the last three months
* Age: 35 to 50 years old for middle-age group, and 65 to 80 years old for elderly group.
* BMI: 20 to 29.9 kg/m2
* Normal glucose tolerance (NGT) for groups Elderly and Middle-age

Exclusion Criteria:

* Use of estrogen, progestogen or systemic corticosteroids.
* Hepatic cirrhosis, renal failure or any clinical condition with impaired insulin sensitivity
* Smoking
* Obesity
* Uncontrolled systemic or debilitating diseases

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult normoglycemic subjects
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Geloneze, MD, PhD, Principal Investigator — LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP)
Locations (1):
- LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP), Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Geloneze B, de Oliveira Mda S, Vasques AC, Novaes FS, Pareja JC, Tambascia MA. Impaired incretin secretion and pancreatic dysfunction with older age and diabetes. Metabolism. 2014 Jul;63(7):922-9. doi: 10.1016/j.metabol.2014.04.004. Epub 2014 Apr 12. PMID 24854384

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process took place at the Laboratory of Investigation on Metabolism and Diabetes - LIMED, located at the Medical School of the State University of Campinas (UNICAMP).
Pre-assignment Details: Cross-sectional study conducted with 24 non-obese patients with normal glucose tolerance. Two groups formed: middle-aged (n=12) and aged(n=12). They were healthy and had no significant illness. None were taking drugs that affect insulin sensitivity/secretion or incretin hormones.
Groups:
- Elderly Normal Glucose Tolerance (NGT): Normoglycemic subjects 65-80 years old
- Middle-age Normal Glucose Tolerance (NGT): Middle-age normoglycemic subjects 35 to 50 years old.
Period: Overall Study
Arm/Group | Elderly Normal Glucose Tolerance (NGT) | Middle-age Normal Glucose Tolerance (NGT)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderly Normal Glucose Tolerance (NGT) | Middle-age Normal Glucose Tolerance (NGT) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 (0) | 0 (0) | 0 (0)
  Between 18 and 65 years | 0 (0) | 12 (0) | 12 (0)
  >=65 years | 12 (0) | 0 (0) | 12 (0)
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (2) | 44 (4) | 54 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Brazil | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Homeostasis Model Assessment Insulin Resistance (HOMA-IR) Index
Description: Insulin sensitivity index calculated as HOMA-IR = (Glucose * Insulin) / 22.5, where glucose is mmol/L and insulin is mili-units (mU)/L. Higher values indicate lower insulin sensitivity.
Time Frame: within 1 month from screening visit
Population: minimum number required to find a significant difference between groups considering the intra-subject variation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elderly Normal Glucose Tolerance (NGT) | Middle-age Normal Glucose Tolerance (NGT)
Number analyzed (Participants) | 12 | 12
units on a scale | 1.91 (1.0) | 0.84 (0.21)
Statistical Analysis 1: Comparison: Elderly Normal Glucose Tolerance (NGT) vs Middle-age Normal Glucose Tolerance (NGT); Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.07

2. Primary Outcome: Glucose Infusion Rate
Description: Whole-body insulin sensitivity, as estimated by the mean glucose infusion rate corrected for fat-free mass(FFM){mg*[kg(FFM)^-1]*min*10} at last 60 min of 180-min hyperglycemic clamp
Time Frame: within 1 month from screening visit
Measure: Mean (Standard Deviation); unit: mg*[kg(FFM)^-1]*min*10
Arm/Group | Elderly Normal Glucose Tolerance (NGT) | Middle-age Normal Glucose Tolerance (NGT)
Number analyzed (Participants) | 12 | 12
mg*[kg(FFM)^-1]*min*10 | 0.48 (0.16) | 1.73 (0.13)
Statistical Analysis 1: Comparison: Elderly Normal Glucose Tolerance (NGT); Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.25

3. Primary Outcome: Adaptive Beta-cell Insulin Production. The Product of Meal Tolerance Test-derived Insulinogenic Index (IGI) for Clamp-derived Insulin Sensitivity Index (ISI) in Normoglycemic Subjects After 65 Years Old in Comparison With Middle-age Normoglycemic Subjects
Description: Beta-cell function was determinated as the beta-cell secretion measured by meal tolerance test adjusted by insulin sensitivity assessed by the hyperglycemic clamp test:Insulinogenic Index/Insulin Sensitivity Index adjusted by free fat mass
Time Frame: within 1 month from screening visit
Measure: Mean (Standard Deviation); unit: (μmol∙kg-1min-1)
Arm/Group | Elderly Normal Glucose Tolerance (NGT) | Middle-age Normal Glucose Tolerance (NGT)
Number analyzed (Participants) | 12 | 12
(μmol∙kg-1min-1) | 1.7 (0.9) | 3.4 (1.3)
Statistical Analysis 1: Comparison: Elderly Normal Glucose Tolerance (NGT) vs Middle-age Normal Glucose Tolerance (NGT); Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Distinctive Beta-cell Function From the Arginine Stimulation Test in Normoglycemic Subjects After Sixty-five Years Old in Comparison With Middle-age Normoglycemic Subjects.
Description: Distinctive beta-cell function as measured by the disposition index - based on the acute insulin response from the arginine stimulation test versus glucose infusion rate adjusted by free fat mass from hyperglycemic clamp - in normoglycemic subjects after sixty-five years old in comparison with middle-age normoglycemic subjects.
Time Frame: within 1 month from screening visit
Measure: Mean (Standard Error); unit: (μmol∙kg-1.min-1)
Arm/Group | Elderly NGT | Middle-age NGT
Number analyzed (Participants) | 12 | 12
(μmol∙kg-1.min-1) | 328.5 (303.4) | 223.5 (174.9)
Statistical Analysis 1: Comparison: Elderly NGT vs Middle-age NGT; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Serum Dipeptidyl Peptidase IV (DPP-IV) Concentration
Description: measured in fasting serum sample by ELISA kit
Time Frame: within 1 month from screening visit
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Elderly Normal Glucose Tolerance (NGT) | Middle-age Normal Glucose Tolerance (NGT)
Number analyzed (Participants) | 12 | 12
pg/ml | 1466.6 (1088.8) | 1458.2 (1006.9)
Statistical Analysis 1: Comparison: Elderly Normal Glucose Tolerance (NGT) vs Middle-age Normal Glucose Tolerance (NGT); Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: GLP-1 Area Under the Curve (AUC)
Description: Area under the curve of glucagon-like peptide (GLP-1) concentrations (measured by ELISA kit) from time 0 to 180 min during a standard meal tolerance test, calculated by the trapezoidal rule.
Time Frame: 1 month from screening visit
Measure: Mean (Standard Deviation); unit: pg/ml/min
Arm/Group | Elderly Normal Glucose Tolerance (NGT) | Middle-age Normal Glucose Tolerance (NGT)
Number analyzed (Participants) | 12 | 12
pg/ml/min | 1061.7 (354.4) | 1027.1 (164.9)
Statistical Analysis 1: Comparison: Elderly Normal Glucose Tolerance (NGT) vs Middle-age Normal Glucose Tolerance (NGT); Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Elderly Normal Glucose Tolerance (NGT) | Middle-age Normal Glucose Tolerance (NGT)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No